CLINICAL TRIAL: NCT01230970
Title: A Phase II, Open-label, Exploratory Study to Assess the Short Term Intratumoural and Peripheral Effects of BN83495 Administered for 14 Days Prior to Surgery to Postmenopausal Women With Newly Diagnosed Primary Invasive Oestrogen Receptor Positive Breast Cancer
Brief Title: Exploratory Study to Assess the Short Term Intratumoural and Peripheral Effects of BN83495 in Postmenopausal Women With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The futility analysis of study NCT00910091 in patients with endometrial cancer shows that the primary endpoint will not be reached.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: X-55-58064-005
Record Dates: First submitted 2010-10-20; First posted 2010-10-29 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — irosustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BN83495 (Experimental): 40mg tablet oral daily administration from Day 1 to Day 14.
  Interventions: Drug: BN83495

INTERVENTIONS:
Drug: BN83495 — 40mg tablet oral daily administration from Day 1 to Day 14.

SUMMARY:
This trial will assess the intratumoural pharmacological activity of BN83495 by changes in intratumoural levels of sex hormones and associated inhibition of steroid sulphatase (STS) activity.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 55 to 80 years with histologically or cytologically documented primary intraductal or lobular invasive breast cancer that meets the following criteria:
* T2, N0 or N1, M0.
* Primary tumour clinically determined to be 2 to 5 cm in the greatest dimension.
* Laboratory documentation of positive oestrogen receptor (ER+) status in at least 10% of the tumour cells.
* Laboratory documentation of HER-2 negative status.

Postmenopausal defined as

* no spontaneous menses for a total of 2 years
* amenorrheic for at least 12 months with serum oestrogen level <30 pg/mL, and both luteinising hormone (LH)/follicle stimulating hormone (FSH) >20 IU/L, chemotherapy-induced amenorrhoea for at least 12 months
* bilateral oophorectomy, or radiation castration and amenorrhoeic for at least 3 months.

Eastern Cooperative Oncology Group (ECOG) performance status ≤2.

Exclusion Criteria:

* Has locally advanced breast cancer that is considered non-operable without neoadjuvant therapy.
* Has evidence of metastatic disease
* as a diagnosis of inflammatory breast cancer
* Has ductal carcinoma in situ

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Intratumoural levels of sex hormones | Baseline and Day 14
Intratumoural steroid sulphatase activity | Baseline and Day 14

SECONDARY OUTCOMES:
Change in the intratumoural Ki67 proliferation index | Baseline and Day 14
Proportion of subjects with a decrease in Ki67 staining ≥50% | Baseline and Day 14
Proportion of subjects with complete cell cycle response, defined as Ki67 staining ≤1% | Baseline and Day 14
Change in Apoptotic Index determined by M30 antibody | Baseline and Day 14
Change in Growth Index (Ki67 proliferation index/M30 apoptotic index) | Baseline and Day 14
Change in steroid sulphatase activity in peripheral blood mononuclear cells (PBMCs). | Baseline and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Akershus University Hospital, Lørenskog, Norway